CLINICAL TRIAL: NCT01018121
Title: LAUNCH II: Learning About Activity and Understanding Nutrition for Better Child Health
Brief Title: Behavioral Rx & Nutrition in Pediatric Chronic Disease
Acronym: LAUNCH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Lori J. Stark Director of Behavioral Medicine and Clinical Psychology, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103254; K24DK059492 (NIH)
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Pediatric Obesity
Keywords: Behavioral Treatment; Preschool Children; Obesity Treatment
MeSH Terms: conditions — Pediatric Obesity | interventions — Spacecraft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinic and Home Behavioral Intervention (Experimental)
  Interventions: Behavioral: LAUNCH
- Pediatrician Counseling (Active Comparator)
  Interventions: Other: Pediatrician Counseling

INTERVENTIONS:
Behavioral: LAUNCH — A 6-month intervention consisting of two phases: Phase I (Intensive Intervention), 12 weekly sessions that alternated between group-based clinic sessions (parent and child concurrent groups) and individual home visits and Phase II (Maintenance), 12 weeks of every other week sessions, alternating between group sessions in-clinic and home sessions. Targeted 3 components: 1) Dietary education with age-specific caloric targets, healthy eating recommendations for children following the AAP guidelines used in the PC session; 2) Physical Activity education with age-specific activities for children and families; and 3) Parenting skills to achieve the diet and physical activity goals using behavioral management skills and parent modeling of eating and activity.
  Arms: Clinic and Home Behavioral Intervention
Other: Pediatrician Counseling — A one time 45-minute visit with a board certified pediatrician for each family that focused on the AAP guidelines for eating and physical activity for children
  Arms: Pediatrician Counseling

SUMMARY:
The objective of this project is to pilot test a behavioral intervention for modifying the diet and physical activity patterns of overweight preschool children through improved parenting and nutritional education(LAUNCH). This intervention will be compared to standard of care for preschool overweight in the primary care setting using a randomized clinical trial design (RCT. The results of this pilot RCT will provide data integral to estimating the effect size for a more definitive RCT of the intervention in the future. The primary hypothesis is:

H1: LAUNCH will result in a significantly greater decrease in BMI z score compared to the standard of care at 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. child age between 2- 5 years;
2. child > 95th percentile BMI for age and sex 12, but not more than 100% above the mean BMI;
3. medical clearance from pediatrician; and
4. at least one parent with a BMI > 25. -

Exclusion Criteria:

1. non-English speaking;
2. living more than 50 miles from the medical center;
3. a disability/illness that would preclude engagement in at least moderate physical activity;
4. medical condition/medication associated with weight gain; or 5) enrolled in another weight control program.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
BMI z score | Baseline, 6 months, 12 months

SECONDARY OUTCOMES:
Parent weight loss | baseline, 24 weeks, 48 weeks
Child caloric intake | baseline, 6 months, 12 months
Home food and activity environment | baseline, 6 months, 12 months
Child physical activity | baseline, 6 motnhs, 12 months
Parent-child mealtime interactions | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori J Stark, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States